CLINICAL TRIAL: NCT05199090
Title: A Randomized, Placebo-controlled, Participant-and-investigator- Blinded, Sponsor Open-label Study to Evaluate the Safety, Tolerability, and Efficacy With Different Dosing Regimens of Subcutaneously Administered MBL949 in Obese Participants With or Without Type 2 Diabetes Mellitus
Brief Title: Study to Assess Safety, Tolerability and Efficacy of SC Administered MBL949 in Obese Participants With or Without T2DM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The tolerability to benefit ratio based on maximum weight loss observed was not considered favorable at the doses studied and the study was terminated early
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CMBL949A12201; 2021-004449-19 (EudraCT Number)
Record Dates: First submitted 2021-12-17; First posted 2022-01-20 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obesity
Keywords: Type 2 diabetes mellitus; weight loss
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MBL949 Arm 1 (Active Comparator): MBL949 one 3 mg dose followed by two doses of 6 mg followed by five doses of 4.5 mg
  Interventions: Drug: MBL949
- MBL949 Arm 2 (Active Comparator): MBL949 two 3 mg doses followed by six doses of 4.5 mg
  Interventions: Drug: MBL949
- MBL949 Arm 3 (Active Comparator): MBL949 one 12 mg dose followed by seven doses of 4.5 mg
  Interventions: Drug: MBL949
- MBL949 Arm 4 (Active Comparator): MBL949 one 1.5 mg dose followed by seven doses of 2.2 mg
  Interventions: Drug: MBL949
- MBL949 Arm 5 (Active Comparator): MBL949 one 3 mg dose followed by two doses of 6 mg followed by five doses of 7.5 mg
  Interventions: Drug: MBL949
- Placebo (Placebo Comparator): Placebo to MBL949
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBL949 — subcutaneous injections administered for 14 weeks
  Arms: MBL949 Arm 1; MBL949 Arm 2; MBL949 Arm 3; MBL949 Arm 4; MBL949 Arm 5
Drug: Placebo — Placebo Comparator to MLB949
  Arms: Placebo

SUMMARY:
This was a multi-center, randomized, placebo-controlled, participant-and-investigator-blinded, sponsor open-label study in obese participants with or without Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The study comprised a screening/baseline period of up to 35 days (5 weeks), a 14-week treatment period in which participants were administered MBL949 or placebo at 8 biweekly intervals starting on Day 1 and a 10-week follow-up period.

Participants were to be enrolled to:

* MBL949 Arm 1, MBL949 Arm 2 and placebo in a 1:1:1 ratio
* MBL949 Arm 3, MBL949 Arm 4 and placebo in a 1:1:1 ratio
* If MBL949 Arm 1 was tolerated, MBL949 Arm 5 was enrolled with a 2:1 ratio (MBL:placebo) within each stratum.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: ≥ 32 kg/m2, weight ≥ 77 kg, stable body weight i.e., less than 1.5 kg self-reported change within 90 days
* Diagnosed T2DM as documented by medical history and confirmed by Investigator and with diagnosed duration < 10 yrs, HbA1c ≤ 9%, and fasting C-peptide ≥ 0.2 ng/ml
* If treated for T2DM, treatment must be limited to diet and exercise and treatment with one of the following anti-diabetic agents (stable for 90 days prior to randomization):

  * Metformin
  * SGLT2i inhibitors (if prescribed as the first line, ie. single agent)
  * DDP4 inhibitors
  * Acarbose

Exclusion Criteria:

* Vitals at screening:

  * systolic blood pressure less than 95 mm Hg or greater than 155 mm Hg
  * diastolic blood pressure less than 60 mg Hg or greater than 95 mm Hg
  * pulse rate less than 56 or greater than 110 bpm
* History of bariatric surgery, Roux-en-Y Gastric Bypass, Sleeve Gastrectomy, gastric banding, and any other intrabdominal procedures designed for weight loss at screening
* History of myocardial infarction with 2 years of screening
* Diet attempts within 90 days before screening
* Participation in organized weight reduction program within 6 months of screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Morehead City, North Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4 research centers in United States participated in the study.
Pre-assignment Details: Participants underwent a screening visit between Day -35 and Day -15 to determine their eligibility for the study.
  On Day 1, participants went to the clinic after an overnight fast of at least 10 hours to complete the Day 1 assessments prior to dosing.
Period: Overall Study
Arm/Group | MBL949 Arm 1 | MBL949 Arm 2 | MBL949 Arm 3 | MBL949 Arm 4 | MBL949 Arm 5 | Placebo
Started | 14 | 22 | 16 | 15 | 15 | 44
Completed | 12 | 8 | 15 | 9 | 10 | 31
Not Completed | 2 | 14 | 1 | 6 | 5 | 13
Not completed — Adverse Event | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 4 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 6 | 0 | 0 | 0 | 5
Not completed — Subject decision | 0 | 4 | 0 | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBL949 Arm 1 | MBL949 Arm 2 | MBL949 Arm 3 | MBL949 Arm 4 | MBL949 Arm 5 | Placebo | Total
Number analyzed (Participants) | 14 | 22 | 16 | 15 | 15 | 44 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (9.53) | 45.8 (7.77) | 44.8 (11.23) | 45.8 (8.98) | 41.6 (10.68) | 44.0 (10.09) | 44.7 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 13 | 12 | 13 | 38 | 101
  Male | 6 | 5 | 3 | 3 | 2 | 6 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 4 | 2 | 6 | 3 | 11 | 29
  White | 11 | 18 | 14 | 9 | 12 | 33 | 97

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Adverse Events
Description: Number of participants with adverse events reported after the first dose of study medication or events present prior to treatment but increase in severity
Time Frame: Baseline to Day 169
Population: Safety Set: included all subjects that received any study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled MBL949: Pooled MBL949 arms
Arm/Group | MBL949 Arm 1 | MBL949 Arm 2 | MBL949 Arm 3 | MBL949 Arm 4 | MBL949 Arm 5 | Pooled MBL949 | Placebo
Number analyzed (Participants) | 14 | 22 | 16 | 15 | 15 | 82 | 44
Participants
  Total AEs | 11 | 20 | 15 | 10 | 14 | 70 | 30
  AEs of mild intensity | 10 | 19 | 15 | 10 | 14 | 68 | 29
  AEs of moderate intensity | 4 | 8 | 7 | 3 | 8 | 30 | 7
  AEs of severe intensity | 0 | 2 | 0 | 1 | 0 | 3 | 2
  Study drug-related AEs | 9 | 18 | 15 | 8 | 12 | 62 | 19
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change-from-baseline in Weight
Description: Baseline weight is defined as the last weight measurement before dosing in kilograms
Time Frame: Week 16
Population: PD analysis set: included all subjects who received any study drug, had Pharmacodynamics (PD) data, and had no protocol deviations with relevant impact on PD data. Only participants with weight data at Baseline and Week 16 were included in the analysis.
Measure: Mean (90% Confidence Interval); unit: kg
Arm/Group | MBL949 Arm 1 | MBL949 Arm 2 | MBL949 Arm 3 | MBL949 Arm 4 | MBL949 Arm 5 | Pooled MBL949 | Placebo
Number analyzed (Participants) | 12 | 8 | 15 | 9 | 10 | 54 | 31
kg | -2.6 [-3.8 to -1.5] | -2.0 [-3.3 to -0.8] | -2.0 [-3.0 to -0.9] | -0.1 [-1.4 to 1.1] | 0.3 [-0.9 to 1.5] | -1.4 [-2.0 to -0.8] | -0.7 [-1.4 to -0.0]
Statistical Analysis 1: Comparison: MBL949 Arm 1 vs Placebo; Comparison of adjusted means; Test type: Other; p = 0.0182, MMRM analysis; adjusted means = -1.9, 80% CI 2-sided [-2.9 to -0.9]
Statistical Analysis 2: Comparison: MBL949 Arm 2 vs Placebo; Test type: Other; p = 0.1205, MMRM analysis; adjusted means = -1.3, 80% CI 2-sided [-2.4 to -0.2]
Statistical Analysis 3: Comparison: MBL949 Arm 3 vs Placebo; Test type: Other; p = 0.0931, MMRM analysis; adjusted means = -1.3, 80% CI 2-sided [-2.2 to -0.3]
Statistical Analysis 4: Comparison: MBL949 Arm 4 vs Placebo; Test type: Other; p = 0.4994, MMRM analysis; adjusted means = 0.6, 80% CI 2-sided [-0.5 to 1.7]
Statistical Analysis 5: Comparison: MBL949 Arm 5 vs Placebo; Test type: Other; p = 0.2295, MMRM analysis; adjusted means = 1.0, 80% CI 2-sided [-0.1 to 2.1]
Statistical Analysis 6: Comparison: Pooled MBL949 vs Placebo; Test type: Other; p = 0.2114, MMRM analysis; adjusted means = -0.7, 80% CI 2-sided [-1.3 to 0.0]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 10 weeks post treatment, up to a maximum duration of 169 days.
Description: Each treatment arm contains a different dosing scheme and adverse event data is provided for the full sequence.
Groups:
- Pooled MBL949: Pooled MBL949
- Total: Total
Arm/Group | MBL949 Arm 1 | MBL949 Arm 2 | MBL949 Arm 3 | MBL949 Arm 4 | MBL949 Arm 5 | Pooled MBL949 | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/22 | 0/16 | 0/15 | 0/15 | 0/82 | 0/44 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/22 | 0/16 | 0/15 | 0/15 | 0/82 | 0/44 | 0/126
Other Adverse Events (participants affected / at risk) | 11/14 | 20/22 | 15/16 | 10/15 | 14/15 | 70/82 | 26/44 | 96/126
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MBL949 Arm 1 (N=14) | MBL949 Arm 2 (N=22) | MBL949 Arm 3 (N=16) | MBL949 Arm 4 (N=15) | MBL949 Arm 5 (N=15) | Pooled MBL949 (N=82) | Placebo (N=44) | Total (N=126)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 3 | 5 | 8
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 2 | 5 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 3
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 5 | 5 | 1 | 2 | 16 | 2 | 18
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 2 | 6 | 5 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 3
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 3
Nausea (Gastrointestinal disorders) | 9 | 17 | 14 | 6 | 12 | 58 | 17 | 75
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 10 | 8 | 6 | 7 | 32 | 3 | 35
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Fatigue (General disorders) | 0 | 5 | 1 | 1 | 1 | 8 | 0 | 8
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Injection site reaction (General disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 2 | 5
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 4 | 1 | 0 | 6 | 6 | 12
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Fungal foot infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 2 | 1 | 3 | 9 | 1 | 10
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 5 | 3 | 8
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Viral infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 4 | 0 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Cortisol free urine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 1 | 5 | 3 | 8
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Food aversion (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 4
Headache (Nervous system disorders) | 3 | 4 | 2 | 2 | 3 | 14 | 1 | 15
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 4 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT05199090/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05199090/SAP_001.pdf